CLINICAL TRIAL: NCT05240742
Title: Persistent Complaints After COVID-19: Epidemiology, Pathophysiology, Prediction, and Communication, the CORona Follow Up (CORFU) Study
Brief Title: CORona (COVID-19) Follow Up Study: Epidemiology, Pathophysiology, Prediction, and Communication
Acronym: CORFU
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); Radboud University Medical Center (Other); Amsterdam University Medical Center (Other); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other)
Responsible Party: Principal Investigator, Sander van Kuijk, Clinical Epidemiologist, Maastricht University Medical Center
Other Study IDs: METC2021-2990
Record Dates: First submitted 2021-11-26; First posted 2022-02-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Long COVID; Post COVID-19 Condition
Keywords: Epidemiology; Pathophysiology; Prediction model; Patient platform
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dutch COVID-19 patients: The study population consists of Dutch (former) COVID-19 patients who have been included in one of the cohorts and categorized in various subgroups:
  * Patients who suffered from (confirmed) COVID-19 and were admitted to the hospital ward.
  * Patient who suffered from (confirmed) COVID-19 and were admitted to the ICU.
  * Patients who suffered from (confirmed or suspected) COVID-19 at home.
  * Patients who suffered from (confirmed) COVID-19 and were in need of inpatient or outpatient rehabilitation after infection at home or in the hospital (ward and/or ICU).
  Interventions: Other: no intervention, the CORFU study conducts analyses based on data which has been prospectively collected (and aggregated when possible) in 7 existing cohorts
- Dutch controls who did not experience COVID-19: One of the cohorts, the POPCOrn cohort, is a community-based cohort which partly consists of controls who did not experience COVID-19
  Interventions: Other: no intervention, the CORFU study conducts analyses based on data which has been prospectively collected (and aggregated when possible) in 7 existing cohorts

INTERVENTIONS:
Other: no intervention, the CORFU study conducts analyses based on data which has been prospectively collected (and aggregated when possible) in 7 existing cohorts — (Clinical) baseline and follow-up data will be collected in the 7 existing cohorts. These data will be aggregated (when possible). The CORFU analyses will be conducted based on the aggregated data.
  Other Names: Integrated database

SUMMARY:
The CORFU study, funded by ZonMW, is a prospective, multiple, cohort study with a maximum follow-up of 24 months after COVID-19. Dutch COVID-19 patients from 7 existing prospective cohorts, aiming and designed to conduct COVID-19 research, will be included in this study.

The CORFU study has 5 aims, divided into 4 work packages (WPs):

1. To describe the nature, severity, pattern and duration of long COVID complaints up to a maximum of two years after infection and its relationship with quality of life (WP1);
2. To describe the rehabilitation and corresponding activities for the treatment and improvement of complaints and quality of life (WP1);
3. To describe the pathophysiological processes that cause long COVID complaints, and the role of vulnerability/resilience factors (WP2);
4. To develop a prediction model for the persistence of complaints, with distinction between patients with and without pre-existing morbidity (WP3);
5. To develop a patient platform prototype in which patients can digitally consult their answers and compare their answers with reference populations (WP4, in collaboration with the EuroQol foundation).

The 7 cohorts participating in the CORFU study are: POPCOrn, COVAS, ELVIS, MaastrICCht, DC&TC, CAPACITY-COVID, and Adelante cohort.

(Clinical) baseline and follow-up data has been collected in these cohorts and will be used/aggregated to investigate CORFU study aims. In addition, questionnaires will be send to the (former) patients of the existing cohorts and patients will be asked about several domains such as persisting complaints and quality of life, at several moments, depending on when the patients have experienced COVID-19. Within this study a patient platform prototype will be developed, together with the EuroQol foundation, to be able to inform patients about the individual situation and course of disease.

ELIGIBILITY:
All 7 existing cohorts have specific inclusion and exclusion criteria.

For the CORFU study, in general, the criteria are:

Patients with proven or suspected COVID-19:

* Confirmed (or suspected) COVID-19 - both home-isolated patients and patients who were admitted to the hospital ward and/or ICU;
* Included in one of the seven cohorts from March 2020 onwards;
* Aged 18 years or older;
* Mastering the Dutch language sufficiently to answer the questionnaires;
* Informed consent.

Controls who did not experience COVID-19:

* Aged 18 years or older;
* Mastering the Dutch language sufficiently to answer the questionnaires;
* Informed consent.

There were no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of Dutch (former) COVID-19 patients and non-COVID-19 controls, who have been included in one of the cohorts and categorized in five subgroups:
  * Patients who suffered from (confirmed) COVID-19 and were admitted to the hospital ward.
  * Patient who suffered from (confirmed) COVID-19 and were admitted to the ICU.
  * Patients who suffered from (confirmed or suspected) COVID-19 at home.
  * Patients who suffered from (confirmed) COVID-19 and were in need of inpatient or outpatient rehabilitation after infection at home or in the hospital (ward and/or ICU).
  * Controls who did not suffer from (confirmed or suspected) COVID-19.
Sampling Method: Probability Sample
Enrollment: 4291 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of long COVID complaints (based on data from all 7 cohorts) | 24 months follow-up after COVID-19
  Long COVID complaints include: exhaustion, respiratory complaints, and mental health complaints.

SECONDARY OUTCOMES:
(Health-related) Quality of life (measured in all 7 cohorts) | 3, 6, 12, 18 and 24 months follow-up after COVID-19
  Measured using the EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) questionnaire. Based on the Dutch tariff, scores range between -0.446 (worst) and 1.000 (best).
Anxiety and depression (measured in all 7 cohorts) | 3, 6, 12, 18 and 24 months follow-up after COVID-19
  Measured using the Hospital Anxiety and Depression Scale (HADS) questionnaire. Scores for both the Anxiety and Depression subscales range from 0 (best) to 21 (worst). A total subscale score of >8 points indicates considerable symptoms of anxiety or depression.
Prevalence of thrombo-embolic complications (not measured in all 7 cohorts) | Measured during COVID-19 hospitalization (baseline), 3, 12, 24 months follow-up after COVID-19
  Thrombo-embolic complications of interest are: acute pulmonary embolism, deep-vein thrombosis, ischemic stroke, myocardial infarction and systemic arterial embolism
  The diagnosis, and therefore, the prevalence of various thrombo-embolic complications will be measured based on a combination of cardiovascular and thrombosis and haemostasis biomarkers (such as troponin I, CK-MB, APTT, and D-dimer), radiologic imaging techniques (computed tomography pulmonary angiography (CTPA), compression ultrasonography (CUS), echocardiography, CT scan of the brain, and CT angiography of the carotid and intracerebral arteries), and electrocardiogram.
Physical functioning (not measured in all 7 cohorts) | Measured during admission in the rehabilitation clinic (baseline), 3, 6, 12 months follow-up
  Measured using the 6 minute walk test (6MWT). The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility. The 6MWT result will be reported as a percentage of the predicted Dutch reference value which is based on the patient's age, sex, length and weight. A score <82% of the predicted value is considered deviant.
Prevalence of cardiovascular diseases (not measured in all 7 cohorts) | Measured during COVID-19 hospitalization (baseline), 1 week, 1 month, and through study completion, an average of 2 years
  Cardiovascular diseases of interest are: coronary artery disease, heart failure, myocardial fibrosis, myocarditis, pericarditis.
  The diagnosis, and therefore, the prevalence of various cardiovascular diseases will be measured based on a combination of radiologic imaging techniques (such as cardiac magnetic resonance, CT and echocardiography), cardial biomarkers (such as troponin and CK-MB), and electrocardiogram.
Prevalence of endothelium dysfunction (not measured in all 7 cohorts) | Measured during COVID-19 hospitalization (baseline), 3, 12 months after COVID-19
  Measured using several biomarkers (such as endothelin-1, coagulation and inflammatory cytokines).
Disease severity during intensive care unit stay (not measured in all 7 cohorts) | Measured on the day of admission with COVID-19 to the intensive care unit (baseline), followed by daily measurement until discharge, an average of 18 days
  Measured using the Sequential Organ Failure Assessment (SOFA) score which is based on the degree of dysfunction of six organ systems. For each organ system, scores range between 0 (best) to 4 (worst). A sum score per day at the intensive care unit can be calculated, which ranges between 0 (best) and 24 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Sander MJ van Kuijk, PhD, Principal Investigator — Maastricht University Medical Center; Chahinda Ghossein-Doha, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nicol B, Rowbotham DJ, Lambert DG. Glutamate uptake is not a major target site for anaesthetic agents. Br J Anaesth. 1995 Jul;75(1):61-5. doi: 10.1093/bja/75.1.61. PMID 7669472
- [Background] Kozlov IA, Piliaeva IE, Matveev IuG, Kormer AIa. [Anesthesiological management in transplantation of the heart after temporary mechanical substitution of its function]. Anesteziol Reanimatol. 1994 Jan-Feb;(1):16-22. Russian. PMID 8010503
- [Background] Keogh JP, Gordon J. Occupational lead poisoning: who should conduct surveillance and training? Am J Ind Med. 1994 Nov;26(5):713-5. doi: 10.1002/ajim.4700260513. PMID 7832218
- [Background] Pittaluga A, Raiteri M. HIV-1 envelope protein gp120 potentiates NMDA-evoked noradrenaline release by a direct action at rat hippocampal and cortical noradrenergic nerve endings. Eur J Neurosci. 1994 Nov 1;6(11):1743-9. doi: 10.1111/j.1460-9568.1994.tb00566.x. PMID 7874313
- [Background] Kaluzewski S, Jagielski M, Rastawicki W, Kochman M. [Evaluation of occurrence of infections caused by Mycoplasma pneumoniae during 1970-1973 based on serological investigations]. Przegl Epidemiol. 1994;48(3):165-72. Polish. PMID 7938618
- [Background] Leijte WT, Wagemaker NMM, van Kraaij TDA, de Kruif MD, Mostard GJM, Leers MPG, Mostard RLM, Buijs J, van Twist DJL. [Mortality and re-admission after hospitalization with COVID-19]. Ned Tijdschr Geneeskd. 2020 Nov 19;164:D5423. Dutch. PMID 33332036
- [Background] Haber J, Wattles J, Crowley M, Mandell R, Joshipura K, Kent RL. Evidence for cigarette smoking as a major risk factor for periodontitis. J Periodontol. 1993 Jan;64(1):16-23. doi: 10.1902/jop.1993.64.1.16. PMID 8426285
- [Background] Skelton-Stroud PN, Glaister JR. Oxalate nephrosis in Macaca fascicularis. Lab Anim. 1994 Jul;28(3):265-9. doi: 10.1258/002367794780681705. PMID 7526030
- [Background] Schwarz T, Sindern S, Bartholmes P, Kaufmann M. The use of a hollow fiber membrane module in sample conditioning prior to electrophoresis. Electrophoresis. 1994 Aug-Sep;15(8-9):1118-9. doi: 10.1002/elps.11501501168. PMID 7859717
- [Derived] Klein DO, Waardenburg SF, Janssen EBNJ, Wintjens MSJN, Imkamp M, Heemskerk SCM, Birnie E, Bonsel GJ, Warle MC, Jacobs LMC, Hemmen B, Verbunt J, van Bussel BCT, van Santen S, Kietelaer BLJH, Jansen G, Klok FA, de Kruif MD, Vernooy K, Haagsma JA, Asselbergs FW, Linschoten M, Cals JWL, Ten Cate H, van der Horst ICC, Wilmes N; CAPACITY-COVID Collaborative Consortium; Ghossein-Doha C, van Kuijk SMJ. Two years and counting: a prospective cohort study on the scope and severity of post-COVID symptoms across diverse patient groups in the Netherlands-insights from the CORFU study. BMJ Open. 2025 Sep 11;15(9):e093639. doi: 10.1136/bmjopen-2024-093639. PMID 40940063
- [Derived] Jacobs LMC, Wintjens MSJN, Nagy M, Willems L, Ten Cate H, Spronk HMH, van Kuijk SMJ, Ghossein-Doha C, Netea MG, Groh LA, van Petersen AS, Warle MC. Biomarkers of sustained systemic inflammation and microvascular dysfunction associated with post-COVID-19 condition symptoms at 24 months after SARS-CoV-2-infection. Front Immunol. 2023 Oct 5;14:1182182. doi: 10.3389/fimmu.2023.1182182. eCollection 2023. PMID 37868959
- [Derived] Ghossein-Doha C, Wintjens MSJN, Janssen EBNJ, Klein D, Heemskerk SCM, Asselbergs FW, Birnie E, Bonsel GJ, van Bussel BCT, Cals JWL, Ten Cate H, Haagsma J, Hemmen B, van der Horst ICC, Kietselaer BLJH, Klok FA, de Kruif MD, Linschoten M, van Santen S, Vernooy K, Willems LH, Westerborg R, Warle M, van Kuijk SMJ. Prevalence, pathophysiology, prediction and health-related quality of life of long COVID: study protocol of the longitudinal multiple cohort CORona Follow Up (CORFU) study. BMJ Open. 2022 Nov 29;12(11):e065142. doi: 10.1136/bmjopen-2022-065142. PMID 36446465
- See also: CAPACITY COVID-19: Registry of patients with COVID-19 including cardiovascular risk and complications — https://capacity-covid.eu/